CLINICAL TRIAL: NCT03226782
Title: Comparison of the Effect of Two Household Physical Exercise Protocols in the Quality of Life and Physical Fitness of Elderly Women With Breast Cancer in Hormoniotherapy Treatment: Interventional Study
Brief Title: Physical Exercise in the Quality of Life and Physical Fitness of Elderly Women With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Professor Fernando Figueira Integral Medicine Institute (Other)
Responsible Party: Principal Investigator, José Roberto da Silva Junior, José Roberto da Silva Junior, Professor Fernando Figueira Integral Medicine Institute
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: U1111-1191-6340
Record Dates: First submitted 2017-07-20; First posted 2017-07-24 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Breast Cancer; Physical Activity; Physical Fitness; Quality of Life
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short intervention protocol (Active Comparator): Will be offered an instructional material that will consist of a routine of 12 exercises to be performed autonomously for range of motion and muscular fitness, using the environmental resources of the home. It will be suggested a daily frequency in the execution of this exercise routine. Also, stimuli and guidelines will be given for the practice of active movement (walking) so that they accumulate at least 10 to 20 minutes of this activity daily. All control and training guidelines for using the manual will be offered through an introductory lecture and subsequent weekly telephone contacts (twice a week). Participants should complete their respective program for a total period of 12 weeks and mark in the manual how often they performed the exercises.
  Interventions: Other: Short intervention protocol
- Long Intervention protocol (Active Comparator): Consisting of 29 exercises to be performed at home. The guideline is to perform each exercise 6 to 8 times in a gentle manner keeping your attention on movement.
  This Manual guides its implementation in a progressive way and at the end it totals about 30 to 45 min of physical exercises per day. All control and training guidelines for use of the manual will be offered through an introductory lecture and subsequent weekly telephone contacts (twice a week). Participants should complete their respective program for a total period of 12 weeks and mark in the manual how often they performed the exercises. Therefore, it guides the implementation of daily walks with cumulative effect.
  Interventions: Other: Long intervention protocol

INTERVENTIONS:
Other: Short intervention protocol — Will be offered an instructional material that will consist of a routine of 12 exercises to be performed autonomously for range of motion and muscular fitness, using the environmental resources of the home. It will be suggested a daily frequency in the execution of this exercise routine. Also, stimuli and guidelines will be given for the practice of active movement (walking) so that they accumulate at least 10 to 20 minutes of this activity daily. All control and training guidelines for using the manual will be offered through an introductory lecture and subsequent weekly telephone contacts (twice a week). Participants should complete their respective program for a total period of 12 weeks and mark in the manual how often they performed the exercises.
  Arms: Short intervention protocol
Other: Long intervention protocol — This Manual guides its implementation in a progressive way and at the end it totals about 30 to 45 min of physical exercises per day. All control and training guidelines for use of the manual will be offered through an introductory lecture and subsequent weekly telephone contacts (twice a week). Participants should complete their respective program for a total period of 12 weeks and mark in the manual how often they performed the exercises. Therefore, it guides the implementation of daily walks with cumulative effect.
  Arms: Long Intervention protocol

SUMMARY:
Among the possibilities of intervention to minimize the effects of cancer treatment, the exercises are efficient in improving the physical fitness and quality of life of the elderly in treatment. The goal is to compare the effects of two home physical exercise protocols on quality of life and physical fitness of elderly people with breast cancer who are in hormone use. A study was carried out at the Institute of Integral Medicine Professor Fernando Figueira (IMIP) within the Professional Master Program in Palliative Care Associated with the Residency Program in Health, which evaluated the effectiveness of a protocol of 29 exercises with walking sessions, performed at home , In the quality of life and physical fitness of the elderly in the treatment of breast cancer. The results of the mentioned research showed that the elderly showed improvement both in quality of life and physical fitness.

In view of the results and the clinical and functional kinetic observation of these patients, the hypothesis was that a shorter intervention protocol, with fewer exercises with fewer repetitions and a lower degree of difficulty can bring results similar to those found, requiring a shorter time In the accomplishment of the exercises, which can favor the adherence to the protocol by the patients, still achieving positive results in their quality of life and physical fitness.

The elderly will undergo evaluations to characterize the sample through questionnaires, the physical fitness assessment will be performed through the Senior Fitness Test (SFT) and anthropometric evaluation before (beginning of the research), in the 6th week and after the 12th week of the research. It will be offered the elderly, instructional material developed for this research - printed manual. It will consist of a routine of 12 exercises to be performed autonomously for range of motion and muscular fitness, using the environmental resources of the home. All control and training guidelines for using the manual will be offered through an introductory lecture and subsequent weekly telephone contacts (twice a week). Participants should complete their respective program for a total period of 12 weeks and mark in the manual how often they performed the exercises. The control group used a protocol with 29 home exercises in a longer manual. The results will be obtained from the statistical package SPSS 10.0 for Windows and a p <0.05 will be accepted.

DETAILED DESCRIPTION:
For the calculation of the sample size, performed in the program Stata 12 version 12, the results presented in the dissertation of Souza Filho and collaborators were considered. The results of the "Raise" test at the end of the study presented a mean of 14.55 ± 3.12 in the intervention group and a mean of 11.16 ± 2.66 in the control group. A 99% power and a type I error of 5% would require 27 patients In each group. Predicting eventual losses, this number was estimated for 33 patients in each group.

The elderly will be considered in two groups, one group will participate in a program of 29 exercises and a second group will participate in a short program with 12 exercises, will be developed according to the following parameters:

Group 1: A manual will be offered, consisting of 29 exercises to be performed at home. The guideline is to perform each exercise 6 to 8 times in a gentle manner keeping your attention on movement. The first 19 exercises were of range of motion:

1. Stretching of buttocks in dorsal decubitus position
2. Trunk side chain elongation in dorsal decubitus
3. Stretching of hip adductors adopting the "butterfly posture"
4. Global mobilization of the spine by adopting the posture of cats
5. Ankle Mobilization
6. Mobilization of the toes
7. Circular ankle mobilization
8. Self-passive ankle mobilization with sitting individual and flexed hip and knee.
9. Mobilization of the thoracic spine in the sitting posture.
10. Trunk side chain elongation in sitting posture
11. Dislocation of scapular girdle
12. Pelvic girdle dissociation
13. Cervical lateral inclination
14. Flexion and cervical extension
15. Cervical rotational movement (global mobilization)
16. Abduction and flexion of the shoulder
17. Internal and external rotation of the shoulder
18. Arms at the front of the body at the shoulder line, the movement consists of performing scapular abduction and lengthening of the flexors at the same time
19. Mobilization of hand and fingers.

    The 10 subsequent exercises are muscular fitness:
20. Sit-up to strengthen mainly of the musculature of the quadriceps and glutes
21. Sits-ups modified
22. Strengthening of pectoral and biceps
23. Strengthening of pectoral and modified biceps
24. Gastrocnemius and soleus strengthening.
25. Gastrocnemius strengthening and modified soleus
26. Exercise of balance and coordination
27. Strengthening of the brachial and iliopsoas triceps
28. Brachial triceps strengthening
29. Brachial triceps strengthening This Manual guides its implementation in a progressive way and at the end it totals about 30 to 45 min of physical exercises per day. All control and training guidelines for use of the manual will be offered through an introductory lecture and subsequent weekly telephone contacts (twice a week). Participants should complete their respective program for a total period of 12 weeks and mark in the manual how often they performed the exercises. Therefore, it guides the implementation of daily walks with cumulative effect.

    Intervention Group: the elderly will be offered, instructional material developed for this research - printed manual. It will consist of a routine of 12 exercises to be performed autonomously for range of motion and muscular fitness, using the environmental resources of the home. It will be suggested a daily frequency in the execution of this exercise routine. Also, stimuli and guidelines will be given for the practice of active movement (walking) so that they accumulate at least 10 to 20 minutes of this activity daily. All control and training guidelines for use of the manual will be offered through an introductory lecture and subsequent weekly telephone contacts (twice a week). Participants should complete their respective program for a total period of 12 weeks and mark in the manual how often they performed the exercises.

    • Procedures related to the production of the instructional manual: a literature review was carried out in the databases BIREME, PUBMED and in websites of organizations of great influence with the theme Physical Activity and Cancer, in specific breast cancer. In addition to interviews and theoretical-practical conceptions of professionals with significant time in the area in question. This stage lasted three months.

    Within this context, the main exercises of amplitude of movement and muscular aptitude were shown in which the realization was easier, reproducible and similar to movements performed within the Activities of Daily Life. From there, the photos of the original manual were reused for their reduced version and served as illustrations for the exercises. This step lasted 15 days.

    During the same period, the researchers conducted the textbook production that provides a brief explanation with simplified language about the importance of adopting physical exercise in patients with breast cancer under treatment and its impact on the quality of life and physical fitness of the patients. Individuals and some guidelines to get into the habit of regular walking.

    After the development process, it was diagrammed to proceed with its printing in reduced version. This step lasted 30 days.

    The elderly will undergo evaluations for characterization of the sample (questionnaires, physical fitness assessment and anthropometric evaluation) before (beginning of the research), in the 6th week and after the 12th week of the research. In addition, in the 6th week, the patient will attend the sector and demonstrate the accomplishment of any manual for possible corrections of movement pattern.

    The collection for characterization of the sample, evaluations and tests, will be performed at the IMIP on days agreed with the elderly soon after signing the TCLE. It will follow the following structuring:

    • Steps: First step: Characterization data of the sample. Anamnesis and questionnaires will be carried out.

    Second stage: Anthropometric evaluation. Measurements of weight, height, BMI and body composition will be performed.

    Third stage: Screening Pre-evaluation of Signs and Symptoms Acute (Annex 5). Measurements of resting blood pressure, resting heart rate, and questioning of possible signs of discomfort will be performed before releasing the patient to perform the assessments and tests for physical fitness. Patients who present an alteration that prevents them from proceeding to the next station will be marked a new date for the same to complete the evaluation procedure, in order to enable participation in the research and avoid any type of risk.

    Fourth stage: Assessment and tests for physical fitness FTS.

    Used tools
    * Functional Evaluation For the variables of functional physical fitness, the Senior Fitness Test (SFT) will be used, in the test and retest regime (minimum interval of 3 and maximum of 8 days between the tests) that is constituted by seven Specific tests that can measure performance in motor functional abilities on a continuous range of wide range, from the condition of greater fragility to the highest degree of functional physical fitness. It assesses the ability to perform functional movements, such as walking, climbing stairs and getting up, as well as checking the muscular fitness, endurance, flexibility and balance of the elderly. It is easy to administer by the evaluators, does not require medical authorization and is very safe. Each item in the test has follow-up performance standards for men and women aged 60-94 years. In addition, the FTS provides reference values in each test item that help identify whether the individual is at risk of loss of mobility.
    * Anthropometric evaluation The following anthropometric data will be collected A) Body weight: body mass measurement using TANITA® electronic balance. B) Stature: greater distance between the vertex and the soil, the individual being in the orthostatic position; C) Perimeter of abdomen: greater abdominal circumference, measured with anthropometric tape; D) Percentage of fat: measure of the relative amount of fat contained in the body. It will be obtained by perimetry.

    E) Lean body mass index: is the ratio of the lean mass to the square of the height.

    F) Body composition shall be measured using bio-impedance

    • Quality of life assessment Quality of life will be assessed using the questionnaire of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire "core" 30 items (EORTC-QLQ-C30) 30, version 3.0. This instrument has 30 questions, consisting of five functional scales: physical, cognitive, emotional, social and role performance; A scale of quality of life and global health; Symptoms of fatigue, pain, nausea, vomiting, dyspnea, lack of appetite, insomnia, constipation and diarrhea and an item that assesses financial difficulties. The possible responses are: no, little, moderately and a lot, scored respectively from 1 to 4. Thus the QLQ-C30 generates a score of 0 to 100 on the functional and symptom scales according to the EORTC score manual. In the functional scale, zero denotes the worst functioning and 100 the best, while the scale of symptoms is the opposite. Being zero with no symptoms and 100 is the maximum of symptoms present.

    All data will be collected by the researcher and other properly trained collaborating professionals who are part of the IMIP Oncology program and IMIP's Postgraduate Program stricto sensu.

    Quality control will be done through a variety of mechanisms: standardized forms and questionnaires, detailed instructions for interviewers and / or evaluators, training of interviewers and evaluators, review of all forms and questionnaires by fieldwork supervisors, repetition of questions Of questions that present inconsistency after review and meetings with all interviewers and / or evaluators whenever questions arise.

    The secondary data that will be used have already been collected and are part of the research by Souza Filho et al.

    After collecting the data, the collection script will be reviewed and then organized and entered into a spreadsheet for statistical analysis. After an exploratory analysis of the data in order to identify if they met normality, using the Kolmogorov Smirnoff test, the statistical characteristics of the sample and the physical fitness variables will be performed. If the comparison is normal distribution, Between the two groups will be performed through the student t test, otherwise the Mann-Withey test will be performed. To evaluate the pre and post in each group will be performed t Student test paired in case of normality or the Wilcoxon test. For the comparison between the different groups, in order to identify the homogeneity between the groups, the equivalence test (Levene test) will be performed. The results will be obtained from the statistical package SPSS 10.0 for Windows and a p <0.05 will be accepted.

ELIGIBILITY:
Inclusion Criteria: • Be between 60 and 74 years old;

* Have a diagnosis of breast cancer, with staging I or II;
* Being in treatment for breast cancer (hormone therapy);

Exclusion Criteria: • Absolute contraindication for performing physical exercises

* Severe depression assessed by the Geriatric Depression Scale
* Malnutrition (degrees I, II and III), detected by the Body Mass Index (BMI), according to WHO criteria.

Ages: 60 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2016-08-15 (Actual); Primary Completion 2017-02-11 (Actual); Study Completion 2017-02-11 (Actual)

PRIMARY OUTCOMES:
Variation in the performance of Lift and Sitting Test | Change from Baseline in Lift and Sitting Test after 6 and 12 weeks
  Test which comprises the Battery Senior Fitness Test (SFT). Evaluates the Lower body strength according to the number of times the individual stood up and sat down in 30 seconds. Characterized as continuous numeric variable
Variation in the performance of Flexion forearm Test | Change from Baseline in Flexion forearm Test and after 6 and 12 weeks
  Test which comprises the Battery Senior Fitness Test (SFT). Evaluates the upper body strength according to the number of push-ups of forearm in 30 seconds. Characterized as continuous numeric variable.
Variation in the performance of Six Minute Walk Test (6MWT) | Change from Baseline in Six Minute Walk Test (6MWT) after 6 and 12 weeks]
  Test which comprises the Battery Senior Fitness Test (SFT). Evaluates aerobic endurance. Total meters walked for 6 minutes walk. Characterized as continuous numeric variable.
Variation in the performance of March Stationary two minutes Test | Change from Baseline in March Stationary two minutes Test after 6 and 12 weeks
  Test which comprises the Battery Senior Fitness Test (SFT). Evaluates aerobic endurance (alternative test). Total double past stationary in 2 minutes. Characterized as continuous numeric variable.
Variation in the performance of Skip and Vir 2.44 meters test | Change from Baseline in Skip and Vir 2.44 meters test after 6 and 12 weeks
  Test which comprises the Battery Senior Fitness Test (SFT). Assesses motor agility and dynamic balance. Evaluates the time in seconds and hundredths in an established path of 2.44 meters on the route to go and return to starting position. Characterized as continuous numerical variable.
Variation in the performance of Sit and Reach Modified test | Change from Baseline in Sit and Reach Modified test (In the Chair) after 6 and 12 weeks
  Test which comprises the Battery Senior Fitness Test (SFT). Evaluates the lower hemisphere flexibility.
  distance in centimeters reached the tip of the middle fingers and the floor in the sitting position.
  Characterized as continuous numerical variable.
Variation in the performance of Flexibility test of the upper limbs | Change from Baseline in Flexibility test of the upper limbs after 6 and 12 weeks
  Test which comprises the Battery Senior Fitness Test (SFT). Evaluates the flexibility of the upper limbs. It measures the distance in centimeters between the tips of the fingers in the back area. Characterized as continuous numeric variable
Variation in the performance of Muscle strength Test | Change from Baseline in Muscle strength Test after 6 and 12 weeks
  Hand Grip Strength Test. Continuous numeric variable: average kilogram-force

SECONDARY OUTCOMES:
Quality of life | Change from Baseline in Quality of life after 12 weeks
  A generic concept reflecting concern with the modification and enhancement of life attributes. Numeric variable: average score from 0 to 100 for 30 issues of questionnaire developed by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30)

CONTACTS AND LOCATIONS:
Overall Officials: JOSE ROBERTO DA SILVA JUNIOR, DOCTORATE, Principal Investigator — Instituto de Medicina Integral Professor Fernando Figueira; ANA CLARA CARVALHO GONÇALVES GUERRA, MASTER, Study Chair — Instituto de Medicina Integral Professor Fernando Figueira

IPD SHARING:
Plan to Share IPD: No